CLINICAL TRIAL: NCT00418145
Title: Oral Megadose Corticosteroid Therapy of Acute Exacerbations of Multiple Sclerosis (OMEGA)
Brief Title: Study to Evaluate Intravenous and Oral Steroids for Multiple Sclerosis Attacks
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low enrollment - data was not analyzed for this study
Sponsor: Fred Lublin (Other)
Collaborators: National Multiple Sclerosis Society (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Fred Lublin, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 01-0781; RG 3363A8
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Multiple Sclerosis
Keywords: Relapsing Forms of Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- megadose oral methylprednisolone (Experimental): 1400 mg qd/5 days
  Interventions: Drug: megadose oral methylprednisolone
- IV methylprednisolone (Experimental): 1000 mg/qd/5 days
  Interventions: Drug: IV methylprednisolone

INTERVENTIONS:
Drug: megadose oral methylprednisolone — 1400 mg qd/5 days
  Arms: megadose oral methylprednisolone
Drug: IV methylprednisolone — 1000 mg/qd/5 days
  Arms: IV methylprednisolone

SUMMARY:
This clinical trial compares the relative efficacy of treating acute exacerbations of relapsing forms of Multiple Sclerosis with equivalent doses of oral and intravenous (IV) methylprednisolone. This is a randomized, blinded, multi-center study.

DETAILED DESCRIPTION:
Intravenous methylprednisolone has been the standard of care for treating acute MS flares. However, the IV administration is cumbersome, inconvenient and expensive. A true comparison of these different approaches has not been undertaken in rigorous fashion. Prior studies have demonstrated the safety of such high doses of oral steroid. For this proposal we employ equivalent oral dosing (1400 mg/day) and compare that to 1000 mg/day IV therapy in patients seen within seven days of an acute exacerbation of MS.

In addition, there are 2 arms to this double-blind, placebo controlled, randomized trial. One arm has an active IV and an oral placebo while the second arm has an IV placebo and an active oral dose. Therefore, each subject will receive an active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 50 years, inclusive.
* Acute symptomatic exacerbation of MS present for great than 24 hours and less than or equal to 7 days at entry with new or worsening symptoms, and with signs referable to the symptoms; in the absence of a fever or active infection.
* Diagnosis of a relapsing form of multiple sclerosis before randomization as determined by Poser or McDonald Criteria.
* Expanded disability status scale (EDSS) score between 2 and 6.5, inclusive at entry.
* Episodes include study neurologist or neuro-ophthalmologist diagnosed: acute optic neuritis, cerebellar, brainstem dysfunction, myelitis, focal cerebral, and/or definitive focal sensory dysfunction.
* New objective clinical finding other than a sensory exacerbation, or bowel/bladder signs alone. Sensory deficits alone will not qualify except for optic neuritis.
* Subjects may continue on their current immunomodulating therapy (such as interferons or glatiramer acetate) throughout the course of the study. Women who become pregnant after the 5-day treatment of steroids should discontinue immunomodulatory treatment.
* Understand and sign written informed consent prior to any testing under this protocol, including screening tests and evaluations that are not considered part of the subject's routine care.

Exclusion Criteria:

* Any patients treated with systemic corticosteroid use within one month of the index episode at screening.
* Prior use of immunosuppressive treatments within 90 days of index episode (mitoxantrone, azathioprine, IVIg) or plasmapheresis.
* Any patient who is pregnant or breastfeeding.
* Unable to perform the Multiple Sclerosis Functional Composite consisting of: Timed 25-Foot Walk, 9-Hole Peg Test, and Paced Auditory Serial Addition Test (3 second).
* Peripheral or cranial neuropathy as sole problem of acute episode.
* History of any significant cardiac, gastrointestinal, hepatic, pulmonary, or renal disease; immune deficiency; or other medical conditions that would preclude corticosteroid therapy.
* Primary Progressive Multiple Sclerosis (PPMS).
* Previous participation in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2003-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Lublin, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (10):
- United States (10):
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - Maimonides Medical Center, Brooklyn, New York
  - The Jacobs Neurological Institute, Buffalo, New York
  - Hospital For Joint Diseases, New York, New York
  - St. Luke's Roosevelt, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - NY Presbyterian Hospital-Cornell University New York, New York, New York
  - University of Rochester, Rochester, New York
  - University of Vermont, Burlington, Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Study Participants: Overall study participants. Data not available separated by arm. Data is also no longer accessible. Data was with biostatistician who no longer has data.
Period: Overall Study
Arm/Group | Total Study Participants
Started | 16
Completed | 10
Not Completed | 6
Not completed — study terminated | 6

BASELINE CHARACTERISTICS:
Population: 16 participants were enrolled into the study. Data not available separated by arm. Data is also no longer accessible. Data was with biostatistician who no longer has data.
Groups:
- Total Study Participants: Overall study participants - Data not available separated by arm. Data is also no longer accessible. Data was with biostatistician who no longer has data.
Arm/Group | Total Study Participants
Number analyzed (Participants) | 16
Age, Customized [Number; unit: participants]
  age 18-29 | 6
  age 30-39 | 3
  age 40-49 | 7
  age 50+ | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Expanded Disability Status Scale (EDSS) Mean Recovery From Day 0 to Day 28.
Description: There is no data analysis for this study
Time Frame: Day 28 and Day 90
Population: Data is also no longer accessible. Data was with biostatistician who no longer has data.
Arm/Group | Megadose Oral Methylprednisolone | IV Methylprednisolone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Clinical Parameters of the Multiple Sclerosis Functional Composite Scale (MSFC) Between Oral and IV Steroid Therapy in Subjects With Relapsing Forms of MS.
Time Frame: Day 28 and day 90
Population: Data is also no longer accessible. Data was with biostatistician who no longer has data.
Arm/Group | Megadose Oral Methylprednisolone | IV Methylprednisolone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Frequency of Relapse Over Time (up to One Year) When Subjects With Relapsing Forms of MS Are Administered One Course of Oral Methylprednisolone Compared to IV Administration.
Time Frame: Day 28 and day 90 and day 365
Population: Data is also no longer accessible. Data was with biostatistician who no longer has data.
Arm/Group | Megadose Oral Methylprednisolone | IV Methylprednisolone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Improvement Using Targeted Neurological Deficits (TND).
Time Frame: Day 28 and day 90
Population: Data is also no longer accessible. Data was with biostatistician who no longer has data.
Arm/Group | Megadose Oral Methylprednisolone | IV Methylprednisolone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Data is also no longer accessible. Data was with biostatistician who no longer has data.
Arm/Group | Megadose Oral Methylprednisolone | IV Methylprednisolone
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The trial was terminated due to difficulties obtaining drug and matching placebo and the inability to meet recruitment. There was no data analysis done for this trial due to low enrollment and data will not be meaningful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes